CLINICAL TRIAL: NCT00373555
Title: Endobronchial Ultrasonography in the Diagnosis of Sarcoidosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Alain Tremblay, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: E-20269
Record Dates: First submitted 2006-09-07; First posted 2006-09-08 (Estimated); Last update posted 2008-10-02 (Estimated); Status verified 2008-08

CONDITIONS: Sarcoidosis; Mediastinal Diseases
Keywords: Sarcoidosis; mediastinal adenopathy; bronchoscopy; Transbronchial needle aspiration; endobronchial ultrasonography
MeSH Terms: conditions — Sarcoidosis; Mediastinal Diseases | interventions — Bronchoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Bronchoscopy

SUMMARY:
Sarcoidosis is a benign, inflammatory condition which will typically involve the lungs and lymph glands in the chest. Diagnosis is often confirmed with bronchoscopic biopsy. A new method of performing bronchoscopic biopsy of lymph glands in the chest has now been developed which uses real-time endobronchial ultrasonography to better locate the lymph glands. While this technique has been proven to be effective in the diagnosis and staging of lung malignancy, its sensitivity for the diagnosis of sarcoidosis is unclear as smaller samples are obtained compared to the standard approach. This study will aim to randomize 50 patients with a clinical suspicion of sarcoidosis to standard biopsy vs. endobronchial ultrasound guided biopsy of the mediastinal lymph glands in order to compare the sensitivity of these tests for sarcoidosis.

DETAILED DESCRIPTION:
Sarcoidosis is a benign, inflammatory condition which will typically involve the lungs and mediastinal lymph nodes. The diagnosis of sarcoidosis is usually confirmed with tissue biopsy, especially if patients in whom treatment with corticosteroids is required. Asymptomatic patients not requiring treatment may not require biopsy, although this is commonly performed because of patient's preference in confirming the diagnosis and concerns about other diagnostic possibilities such as lymphoma.

Given the predilection of this disease to the chest, the lung and mediastinal lymph nodes are the most common sites for biopsy. Bronchoscopic samples are often obtained initially given their good sensitivity for this disease and low complication rates. If the diagnosis of sarcoidosis is not confirmed by bronchoscopy, more invasive surgical procedures such as mediastinoscopy or open lung biopsy may be required. As such, any improvement in the minimally invasive methods for diagnosis of this condition would be of benefit these patients and may also lead to cost efficiencies for the health care system.

Transbronchial needle aspiration (TBNA) with a 19 gauge "histology" needle has been the standard bronchoscopic approach to the biopsy of mediastinal lymph nodes in patients with suspected sarcoidosis. Using anatomical landmarks and computed tomography (CT) images, the TBNA needle is advanced "blindly" through the airway wall, and into the mediastinal lymph node. Because of the lack of real-time visual guidance, it is possible to miss the targeted lymph node as well as enter vascular structures with the needle system and cause bleeding.

A new method of performing TBNA has now been developed which uses real-time endobronchial ultrasonography to advance a 22 gauge needle into mediastinal lymph nodes under direct visualization (EBUS-TBNA). While this technique has been proven to be effective in the diagnosis and staging of lung malignancy, its sensitivity for the diagnosis of sarcoidosis is unclear given that larger biopsy samples are often required to make this diagnosis.

This study will aim to randomize patients with a clinical suspicion of sarcoidosis and mediastinal adenopathy undergoing bronchoscopy to TBNA vs. EBUS-TBNA in order to compare the sensitivity of these tests for sarcoidosis.

ELIGIBILITY:
Inclusion Criteria:

* age over 16 years
* pathological mediastinal or hilar adenopathy (over 1 cm short axis) confirmed on Computed Tomography (CT) of the chest
* clinical/radiological diagnosis of sarcoidosis is considered likely diagnosis
* clinical decision made by patient and treating physician to proceed to bronchoscopy

Exclusion Criteria:

* absence of informed consent
* uncorrected coagulopathy
* platelets under 100
* INR over 1.3
* use of clopidogrel in the 7 days prior to bronchoscopy
* medical contraindication to bronchoscopy

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2006-09; Primary Completion 2007-09 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield

SECONDARY OUTCOMES:
Sensitivity and specificity for Sarcoidosis
Complication rates
Length of Procedure
Dose of sedation required

CONTACTS AND LOCATIONS:
Overall Officials: Alain Tremblay, MDCM, Principal Investigator — University of Calgary
Locations (1):
- Health Sciences Centre, Calgary, Alberta, Canada

REFERENCES:
- [Derived] Tremblay A, Stather DR, MacEachern P, Khalil M, Field SK. A randomized controlled trial of standard vs endobronchial ultrasonography-guided transbronchial needle aspiration in patients with suspected sarcoidosis. Chest. 2009 Aug;136(2):340-346. doi: 10.1378/chest.08-2768. Epub 2009 Feb 2. PMID 19188547